CLINICAL TRIAL: NCT04524806
Title: Influence of Stabilization Splint Thickness on The Temporomandibular Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: halenurbilir
Record Dates: First submitted 2020-08-16; First posted 2020-08-24 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Temporomandibular Disorder; Temporomandibular Joint Disorders; Orofacial Pain
Keywords: stabilization splint; temporomandibular disorders; RDC/TMD; temporomandibular joint; orofacial pain
MeSH Terms: conditions — Temporomandibular Joint Disorders; Facial Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2 mm-thick splint group (2 mm-TSG) (Active Comparator): The group which applied the 2 mm thick stabilization splint
  Interventions: Other: stabilization splint
- 4 mm-thick splint group (4 mm-TSG) (Active Comparator): The group which applied the 4 mm thick stabilization splint
  Interventions: Other: stabilization splint

INTERVENTIONS:
Other: stabilization splint — Stabilization splint is an appliance which applied to upper or lower jaw and regulating the occlusal forces in the temporomandibular joint that can cause disorders, also preventing excessive contraction of the masticatory muscles

SUMMARY:
The aim of the study is assessing the effect of the stabilization splint (SS) thickness on the temporomandibular disorder's and their symptoms; such as muscle or temporomandibular joint (TMJ) pain, TMJ sounds, and limitation of mouth opening.

DETAILED DESCRIPTION:
Participants are selected from patients who applied to the clinic with the complaint of temporomandibular disorders (TMDs). Symptoms are evaluated with RDC/TMD forms. Regarding the treatment plan, patients are divided into two groups; 2 mm-thick splint group (2 mm-TSG) and 4 mm-thick splint group (4 mm-TSG). They used SS's at night for 8 hours, and they were recalled on 1st, 2nd, 3rd, and 6th months after splint insertion. Their symptoms and splints are checked.

ELIGIBILITY:
Inclusion Criteria:

* No need for orthodontic treatment
* Maximum 2 teeth have been extracted
* Having efficient occlusal contacts
* Patients in the axis 1 and axis 2 groups according to Research Diagnostic Criteria for Temporomandibular Disorders (RDC/TMD)

Exclusion Criteria:

* Treated with stabilization splint before
* Partial edentulous patients
* Patients in the axis 3 group according to Research Diagnostic Criteria for Temporomandibular Disorders (RDC/TMD)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2013-07-01 (Actual); Primary Completion 2014-01-01 (Actual); Study Completion 2015-01-30 (Actual)

PRIMARY OUTCOMES:
Presence of myofascial pain | Up to 6 months
  Myofascial pain and myofascial pain with limited opening are in the Group I according to the RDC/TMD.
  I.a Myofascial pain:
  1. Reported pain in masticatory muscles (In the jaw, temples, face, preauricular area, or inside the ear, at rest or function)
  2. Pain on palpation in at least 3 sites (There are 20 sites (ten on each side): posterior, middle and anterior Temporalis; origin, body and insertion of Masseter; posterior mandibular region; Submandibular region; lateral Pterygoid; tendon of Temporalis), one of them at least in the same side of the reported pain
  I.b Myofascial pain with limited opening:
  1. Myofascial pain
  2. Pain-free unassisted 3 opening< 40 mm and Passive 4 stretch ≥ 5 mm
Presence of intra-capsular temporomandibular disorders | Up to 6 months
  II.a Disc displacement with reduction:
  1. No pain in the joint
  2. Reproducible (All clicks must be reproduced 2 out of 3 consecutive trials) click on excursion with either opening or closing click
  3. With click on opening and closing (unless excursive click confirmed):
     * Click on opening occurs at ≥ 5 mm interincisal distance than on closing
     * Clicks eliminated by protrusive opening
  II.b Disc displacement without reduction with limited opening:
  1. History of locking or catching that interfered with eating
  2. Absence of TMJ clicking
  3. Unassisted opening (even painful) ≤ 35mm and passive stretch ≤ 4mm
  4. Contralateral excursion < 7mm
  II.c Disc displacement without reduction without limited opening:
  1. History of locking or catching that interfered with eating
  2. The presence of TMJ sounds excluding DDR clicking
  3. Unassisted opening (even painful) > 35mm and passive stretch > 4mm
  4. Contralateral excursion ≥ 7mm

SECONDARY OUTCOMES:
Presence of TMJ sounds | Up to 6 months
  Click: A distinct sound, of brief and very limited duration, with a clear beginning and end, which usually sounds like a "click."
  Opening Click: If upon opening and closing from maximum intercuspation, a click is noted on two of three opening movements, record as positive for opening click.
  Closing Click: A click present on two of three closing mandibular movements.
Limitation of jaw movements | Up to 6 months
  The researcher places the edge of the millimeter ruler at the incisal edge of the maxillary central incisor that is the most vertically oriented and measures vertically to the labioincisal edge of the opposing mandibular incisor; records this measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Halenur Bilir, DDS, Study Director — Medipol University; Hanefi Kurt, PhD, Study Chair — Medipol University

IPD SHARING:
Plan to Share IPD: No